CLINICAL TRIAL: NCT03527472
Title: A Randomized Placebo-controlled, Double Blind Phase 2 Clinical Trial of Memantine for the Treatment of Cognitive Impairment in Systemic Lupus Erythematosus
Brief Title: Memantine for the Treatment of Cognitive Impairment in Systemic Lupus Erythematosus
Acronym: ClearMEMory
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Evergreen Therapeutics, Inc. (Industry); The University of Texas Health Science Center, Houston (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, James C. Jackson, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 180256
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: cognitive dysfunction; memantine; lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Cognitive Dysfunction | interventions — Memantine

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Memantine (Experimental): At randomization, subjects will receive 5 mg twice per day for one week. They will escalate their dose to 10 mg twice per day for one week, then 10 mg in the morning and 20 mg at night for one week, and finally 20 mg twice per day for three weeks. Maximum tolerated will be determined at this time and this dose will be continued for an additional six weeks.
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): At randomization, subjects will receive one matching placebo capsule twice per day for one week. They will also take one matching placebo capsule twice per day for the next week (week 2), then one matching placebo capsule in the morning and two capsules at night for one week (week three), and finally two capsules twice per day for three weeks (weeks 4-6). Maximum tolerated number of capsules will be determined at this time and this dose will be continued for an additional six weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Memantine is an FDA-approved drug for the treatment of Alzheimer's disease.
  Other Names: Namenda
  Arms: Memantine
Drug: Placebo — The placebo will match the study drug in appearance, dose, and frequency. It will not contain any active drug (memantine).
  Arms: Placebo

SUMMARY:
A phenome-wide association study (PheWAS) identified an association between a variant in the human gene for the N2A subunit of the N-methyl-D-aspartate (NMDA) receptor, GRIN2A, and Systemic Lupus Erythematosus (SLE). A single nucleotide polymorphism (SNP) in this gene encodes for increased NMDA receptor activity. Based on the potential function of the associated SNP and published literature, alterations in SNP function signaling may underlie a cluster of symptoms. The objective of this study is to evaluate the safety, tolerability and efficacy of memantine, an NMDA receptor antagonist, in a precise patient subset with SLE. Participants will complete a full 14-week clinical trial, receiving either memantine or a placebo. Participants' blood will be drawn to test for various antibodies as well as organ function. Patients' urine will also be collected to assess organ function and pregnancy for females at a number of specific time points. The overall goal is to develop a safe and inexpensive therapeutic approach to reduce debilitating cognitive symptoms in a precisely selected SLE sub-population.

ELIGIBILITY:
Inclusion Criteria:

1. Meet American College of Rheumatology (ACR) criteria for SLE
2. Report NPSLE symptoms on the screening survey recommended by EULAR guideline but limited to the psychiatric manifestations questions
3. Score ≤ 85 on the RBANS total index (≤ 1 SD below the normative mean of 100)

Exclusion Criteria:

1. Male and female subjects <18 or >60 years
2. Change in medication that may affect mood or cognition including prednisone, antidepressant medications, or stimulants within the last 4 weeks
3. Regular (daily) use of opioids or other drugs of abuse including heavy alcohol or marijuana use
4. Metabolic derangement defined as liver function tests >3x upper limit of normal or severe renal disease defined as calculated creatinine clearance <30 mL
5. Severe psychiatric disease including schizophrenia, psychosis, suicidal depression
6. Other factors which in the opinion of the investigator could potentially impact the study outcomes (e.g., underlying disease, medications, history)* or prevent the participant from completing the protocol (poor compliance or unpredictable schedule)
7. Inability or refusal to give informed consent for any reason including a diagnosis of dementia or significant cognitive impairment**
8. Patients who are pregnant
9. Patients who are enrolled in other investigational drug studies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Repeatable Battery for Assessment of Neuropsychological Status (RBANS) Total Index Score at endpoint (Visit 4) | 12 weeks
  RBANS is a widely used psychiatric tool that objectively measures cognitive impairment. It is comprised of 12 subtests and takes approximately 30 minutes. For scoring, the RBANS index scores are converted to classifications including Very Superior (130 and above), Superior (120-129), High Average (110-119), Average (90-109), Low Average (80-89), Borderline (70-79), and Extremely Low (69 and below). A score of Extremely Low equates to severe cognitive impairment. The primary outcome measure will be analyzed using ANCOVA controlling for memantine/placebo, baseline RBANS, sex, age, and NMDAR status.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 weeks
  We will determine the safety of memantine as measured by treatment-emergent adverse events.
Polysymptomatic Distress Scale | 12 weeks
  The Polysymptomatic Distress (PSD) scale measures the effect of PSD over a range of pain-related clinical symptoms. The scale was derived from variables used in the 2010 American College of Rheumatology fibromyalgia criteria, modified for use in clinical research, and broadened to be applicable for patients not meeting fibromyalgia diagnostic criteria. The PSD score is calculated by summing two components, the Widespread Pain Index (WPI) and Symptom Severity Scale (SSS). The WPI is a count of painful nonarticular body regions, and the SSS is a symptom severity measure that includes fatigue, sleep, and cognitive problems.
Beck Depression Inventory | 12 weeks
  The Beck Depression Inventory (BDI) is a 21-item, self-report inventory that measures depression symptoms and attitudes. It takes approximately 10 minutes to complete and requires a fifth to sixth grade reading level to adequately comprehend the questions.
Hospital Anxiety and Depression Scale | 12 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessment scale and was developed to detect states of depression, anxiety, and emotional distress among patients who were being treated for a variety of clinical problems. The scale has a total of 14 items, with responses being scored on a scale of 0-3 (3 indicates higher symptom frequencies). Scores for each subscale (anxiety and depression) range from 0 to 21, categorized as follows: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21.
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)-2K | 12 weeks
  SLEDAI-2K is an updated version of the SLEDAI which was originally developed in 1985 as a clinical index to assess lupus disease activity in the preceding 10 days. It is a cumulative and weighted index of 24 different clinical and laboratory variables/disease descriptors, comprising 9 organ systems. The Investigator will assess disease descriptors on the SLEDAI-2K collection sheet (e.g., arthritis, myositis, alopecia, rash, mucosal ulcers, etc.).
Patient Global Impression of Change | Endpoint (Visit 4)
  Participants will answer the standard question, "Considering all the ways your health affects you, how are you doing since the beginning of your treatment?" Answers include very much worse, much worse, worse, unchanged, improved, much improved, and very much improved.
RBANS Subscales | 12 weeks
  Our primary outcome is the RBANS Total Index Score, which is the sum of several subscales/tests. For a secondary outcome, we will look at each subscale/test individually to see if there is a trend for any one test in particular. The subscales are all scored the same (40 - 160) and include immediate memory, delayed memory, visuospatial/constructional, language, and attention.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie J Crofford, MD, Principal Investigator — Professor of Medicine - Rheumatology
Locations (3):
- United States (3):
  - The Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Health Science Center, Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03527472/ICF_000.pdf